CLINICAL TRIAL: NCT06903429
Title: A Comparative Study to Evaluate Targeting Methods for Axillary Surgery in Patients With Clinically Node-positive Breast Cancer: A Prospective Multicenter Pilot Study
Brief Title: Using LUminoMark vs Coventional Practice for Targeted Axillary Surgery
Acronym: LUCAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Collaborators: Samsung Medical Center (Other); Gangnam Severance Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Myongji Hospital (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, JeeYeon Lee, Associate professor, Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG 36
Record Dates: First submitted 2025-03-11; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Axillary Lymph Nodes; Target Lesion
Keywords: Targeting; Axillary lymph node; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Erythema Multiforme

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LuminoMarkTM group (Experimental): LuminoMarkTM using group for targeting of axillary lymph node
  Interventions: Procedure: Targeting of axillary lymph nodes using LuminoMark
- Conventional group (Active Comparator): Conventional method using group for targeting of axillary lymph node
  Interventions: Procedure: Targeting of axillary lymph nodes using conventional method

INTERVENTIONS:
Procedure: Targeting of axillary lymph nodes using LuminoMark — This group used LuminoMark as a targeting method for axillary lymph nodes in breast cancer patients with suspected metastasis, comparing it to existing methods (charcoal staining, needle targeting, ultrasound-guided skin marking) to assess its safety and effectiveness, with procedural differences based on neoadjuvant chemotherapy status.
  Arms: LuminoMarkTM group
Procedure: Targeting of axillary lymph nodes using conventional method — This group used conventional method (charcoal staining, needle targeting, ultrasound-guided skin marking) as a targeting method for axillary lymph nodes in breast cancer patients with suspected metastasis, with procedural differences based on neoadjuvant chemotherapy status.
  Arms: Conventional group

SUMMARY:
The purpose of this study was to compare the use of LuminoMarkTM as a method of targeting axillary lymph nodes with other existing methods used in each institution, such as charcoal staining, needle targeting, and ultrasound-guided skin marking, in patients with breast cancer clinically suspected of metastasis, with or without clipping at the time of diagnosis, regardless of the presence or absence of neoadjuvant chemotherapy. By doing so, the investigators aimed to confirm the safety and usefulness of LuminoMarkTM as a targeting method.

DETAILED DESCRIPTION:
In breast cancer patients, lymph node targeting plays an important role in determining the stage and setting the treatment policy, and the existing methods for this purpose include charcoal staining, needle targeting, and ultrasound-guided skin marking. However, these methods have limitations in terms of detection rate and accuracy, and a new targeting method, LuminoMarkTM, shows the potential to replace them. The purpose of this study is to evaluate the detection rate and safety of lymph node targeting using LuminoMarkTM in breast cancer patients and to verify its effectiveness by comparing it with existing targeting methods. The study was designed as a prospective comparative study, and patients diagnosed with breast cancer and requiring lymph node targeting were divided into the LuminoMarkTM group and the existing method group. The existing method group selects a standard method among charcoal staining, needle targeting, and ultrasound-guided skin marking to perform targeting, and the lymph node detection rate, procedure time, complication rate, and patient satisfaction are the main evaluation indicators in both groups. After targeting, the suitability of the detected lymph nodes is confirmed through pathological analysis, and appropriate statistical analysis is performed to compare the difference in detection rates of each method. Through this study, the investigators evaluate whether LuminoMarkTM provides superior detection rates and safety compared to existing lymph node targeting methods, and based on this, the investigators aim to suggest a more effective and reliable targeting method for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 70 years
* Women diagnosed with primary invasive breast cancer through biopsy
* Patients with clinically and imaging-suspected axillary lymph node metastasis, confirmed pathologically (aspiration cytology or needle biopsy)
* Clinically staged T1-T4, N1-3
* Patients who have fully understood the clinical trial content (if possible) and signed the informed consent form

Exclusion Criteria:

* Patients with inadequate radiological evaluation of the axilla before surgery
* Recurrent breast cancer or inflammatory breast cancer
* Breast cancer with distant metastasis (Stage 4)
* Patients with a history of hypersensitivity to the components of the investigational drug
* Patients scheduled for axillary dissection that does not require targeting of the target lesion
* Patients with active connective tissue disease (e.g., scleroderma, lupus) that has invaded the skin
* Patients with locally advanced breast cancer or inflammatory locally advanced breast cancer that is not amenable to surgery
* Patients with a history of hypersensitivity to the main component or excipients of the investigational drug
* Female subjects who may become pregnant during the clinical trial period and do not agree to use a highly effective non-hormonal contraception method (e.g., sterilization, intrauterine device, complete abstinence, vasectomy partner) from the time of investigational drug injection until the follow-up visit
* Pregnant or lactating women
* Patients who have participated in another clinical trial within 12 weeks before enrollment in this clinical trial
* Patients deemed unsuitable for participation by the investigator for any other reason

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the axillary lymph node targeting method | From enrollment to the end of observation at 3 weeks
  The outcome will be assessed by determining whether the preoperatively marked (targeted) lymph node is successfully identified and retrieved during surgery, and confirmed by postoperative pathological examination.
  Success (match): The retrieved lymph node is matched with targeted lymph node.
  Failure (not match): The retrieved lymph node is not matched with targeted lymph node.
Comparison the accuracy rate between LuminoMark group and conventional group | At the end of the trial (up to 1 year)
  Compare the rate at which the lymph nodes are accurately detected using charcoal staining, needle targeting, ultrasound-guided marking, etc., with the rate at which they are detected using LuminoMark.

SECONDARY OUTCOMES:
Comparion of surgical time between two group | During surgery
  Comparison of time from skin incision to detection of marked axillary lymph nodes Comparison of total axillary surgical time
Comparison of complications between two groups | From enrollment to the end of observation at 3 weeks
  Compare the postoperative complications after surgery
Adverse drug reactions | From enrollment to the end of observation at 3 weeks
  Compare the incidence of adverse drug reactions between two groups
Concordance rate between sentinel lymph node and targeted lymph node in both group | From enrollment to the end of observation at 3 weeks
  Concordance rate between sentinel lymph node and targeted lymph node in both group

CONTACTS AND LOCATIONS:
Overall Officials: Korean Breast Cancer Society Study Group, Study Director — Korean Breast Cancer Society Study Group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takemoto N, Koyanagi A, Yasuda M, Yamamoto H. Comparison of the indocyanine green dye method versus the combined method of indigo carmine blue dye with indocyanine green fluorescence imaging for sentinel lymph node biopsy in breast conservative therapy for stage </=IIA breast cancer. BMC Womens Health. 2018 Sep 18;18(1):151. doi: 10.1186/s12905-018-0646-5. PMID 30227837
- [Background] Lee J, Kang B, Jung JH, Kim HJ, Kim WH, Yang JD, Lee JS, Chae YS, Lee SJ, Lee IH, Park JY, Park NJ, Park HY. Feasibility of an indocyanine green-hyaluronic acid mixture (LuminoMark) for targeting suspicious axillary lymph nodes in patients with breast cancer. BMC Cancer. 2024 Dec 30;24(1):1588. doi: 10.1186/s12885-024-13175-9. PMID 39736609
- [Background] Bang YJ, Choi HJ, Kim I, Lee MH, Lee S, Shin HJ, Nam SJ, Lee JE, Chae BJ, Lee SK, Ryu JM, Kim SW. The efficacy and safety of an indocyanine green-hyaluronic acid mixture (LuminoMark) for localization in patients with non-palpable breast lesions: A multicenter, randomized, open-label, parallel phase 3 clinical trial. Front Oncol. 2023 Mar 24;13:1039670. doi: 10.3389/fonc.2023.1039670. eCollection 2023. PMID 37035212
- [Background] Kitzman JV, Martin JF, Holley JH, Huber WG. Determination of antipyrine in catfish plasma by high-performance liquid chromatography. J Chromatogr. 1988 Mar 11;437(1):306-10. doi: 10.1016/s0021-9673(00)90399-6. No abstract available. PMID 3372671
- [Background] Lin J, Lin LS, Chen DR, Lin KJ, Wang YF, Chang YJ. Indocyanine green fluorescence method for sentinel lymph node biopsy in breast cancer. Asian J Surg. 2020 Dec;43(12):1149-1153. doi: 10.1016/j.asjsur.2020.02.003. Epub 2020 Mar 3. PMID 32143963
- [Background] White KP, Sinagra D, Dip F, Rosenthal RJ, Mueller EA, Lo Menzo E, Rancati A. Indocyanine green fluorescence versus blue dye, technetium-99M, and the dual-marker combination of technetium-99M + blue dye for sentinel lymph node detection in early breast cancer-meta-analysis including consistency analysis. Surgery. 2024 Apr;175(4):963-973. doi: 10.1016/j.surg.2023.10.021. Epub 2023 Dec 13. PMID 38097484
- [Background] Bargon CA, Huibers A, Young-Afat DA, Jansen BAM, Borel-Rinkes IHM, Lavalaye J, van Slooten HJ, Verkooijen HM, van Swol CFP, Doeksen A. Sentinel Lymph Node Mapping in Breast Cancer Patients Through Fluorescent Imaging Using Indocyanine Green: The INFLUENCE Trial. Ann Surg. 2022 Nov 1;276(5):913-920. doi: 10.1097/SLA.0000000000005633. Epub 2022 Jul 27. PMID 35894448
- [Background] Kim WH, Kim HJ, Jung JH, Park HY, Lee J, Kim WW, Park JY, Chae YS, Lee SJ. Ultrasound-Guided Restaging and Localization of Axillary Lymph Nodes After Neoadjuvant Chemotherapy for Guidance of Axillary Surgery in Breast Cancer Patients: Experience with Activated Charcoal. Ann Surg Oncol. 2018 Feb;25(2):494-500. doi: 10.1245/s10434-017-6250-3. Epub 2017 Nov 13. PMID 29134374
- [Background] Kim WH, Kim HJ, Jung JH, Park HY, Lee J, Kim WW, Park JY, Cheon H, Lee SM, Cho SH, Shin KM, Kim GC. Ultrasound-Guided Fine-Needle Aspiration of Non-palpable and Suspicious Axillary Lymph Nodes with Subsequent Removal after Tattooing: False-Negative Results and Concordance with Sentinel Lymph Nodes. Ultrasound Med Biol. 2017 Nov;43(11):2576-2581. doi: 10.1016/j.ultrasmedbio.2017.07.011. Epub 2017 Aug 19. PMID 28830644
- [Background] Lee J, Jung JH, Kim WW, Lee RK, Kim HJ, Kim WH, Park JY, Jeong JY, Chae YS, Lee SJ, Park SH, Kim MY, Yang JD, Lee JW, Lee JS, Park HY. 5-year oncological outcomes of targeted axillary sampling in pT1-2N1 breast cancer. Asian J Surg. 2019 Jun;42(6):681-687. doi: 10.1016/j.asjsur.2018.10.004. Epub 2018 Nov 22. PMID 30470459